CLINICAL TRIAL: NCT07069803
Title: Long-term Oncologic Outcomes of Minimal Access (Endoscopic or Robotic Assisted) Nipple-sparing Mastectomy Compared With Conventional Approach in Breast Cancer - a Propensity Score Matching Analysis
Brief Title: Oncologic Outcomes of Minimal Access Nipple-sparing Mastectomy Compared With Conventional Approach in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CCH-IRB-231217
Record Dates: First submitted 2025-06-26; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: nipple-sparing mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- minimal acccess NSM: minimal acccess NSM
- conventional NSM: conventional NSM

SUMMARY:
In this study the investigators investigate the oncological outcomes of minimal access nipple sparing mastectomy compared with conventional nipple sparing mastectomy for the treatment of breast cancer

DETAILED DESCRIPTION:
A retrospective analysis of a prospectively collected database was conducted from single institute to compare the oncologic outcomes of MA-NSM versus C-NSM. The clinical results and oncologic outcome (margin involved rate, local recurrence and overall survival) were compared between groups. To prevent bias, a case control approach was conducted with propensity score matching (PSM) method.

ELIGIBILITY:
Inclusion Criteria:

* primary operable breast cancer and had undergone NSM

Exclusion Criteria:

* had metastatic disease, non-malignant breast disease cases, bilateral breast cancer cases, recurrent breast cancer as well as male breast cancer cases and patients who did not undergo NSM

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSM patients at CCH
Sampling Method: Probability Sample
Enrollment: 1129 (Actual)
Dates: Start 2000-02-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
local recurrence | 10 years
  local recurrence
distant metastasis | 10 years
  distant metastasis
disease free survival | 10 years
  disease free survival
overall survival | 10 years
  overall survival

SECONDARY OUTCOMES:
operative duration | during surgery
  operative duration
intra-operative blood loss | during surgery
  intra-operative blood loss
post-operative complications | 30 days post-operatively
  post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Jun Su, MBBS, FRCS, Study Director — Changhua Christian Hospital